CLINICAL TRIAL: NCT00682695
Title: Genetic and Environmental Risk Factors for Hemorrhagic Stroke
Acronym: GERFHS
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Maryland, Baltimore (Other); Massachusetts General Hospital (Other); Duke University, Durham, NC (Unknown); Columbia University (Other); University of Illinois at Chicago (Other); Baptist Health, Louisville (Other)
Responsible Party: Principal Investigator, Daniel Woo, Professor, State University of New York at Buffalo
Other Study IDs: NS36695; 2U01NS036695-15A1 (NIH)
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: stroke; brain attack; hemorrhagic stroke; risk factors
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood DNA, RNA and Complete Blood Count (CBC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants who have had a hemorrhagic stroke at University of Maryland, University of Cincinnati, Massachusetts General Hospital, Duke University, Columbia University and University of Chicago Illinois, age 18 years or greater. Ability of the patient or legal representative to provide informed consent. Racial/ethnic category meets one of the following: African American, Caucasian or Hispanic.
  Healthy volunteers who are matched to the study cases with hemorrhagic stroke within +/- 5 years of age, same gender and same race.

SUMMARY:
The purpose of this study is to find risk factors for hemorrhagic stroke.

DETAILED DESCRIPTION:
The proposed research builds on the most robust, statistically significant and replicated association identified to determine the mechanism by which it may relate to intracerebral hemorrhage (ICH) risk. Given that ICH is an extreme phenotype on a spectrum of manifestations of cerebral small vessel disease, the findings that emerge from our proposed studies offer the promise of broad impact for research and treatment in a wide variety of cerebrovascular disorders.

In the genetic epidemiology of hemorrhagic stroke, we propose to perform an in-depth fine-mapping of the entire 1q22 genomic region (~250kb) to investigate whether genetic variants influence gene expression that correlates with ICH status or changes in expression over time in ICH cases. As existing samples were not processed for gene expression analysis, we will recruit 500 non-lobar ICH cases (~150 black, ~350 white) and 1000 controls (300 black, 700 white) to correlate sequence variation with gene expression levels in the same samples. Identified associations will be replicated in 6,000 cases of ICH and 9,361 individuals in the CHARGE consortium with MRI white matter hyperintensity volume measurements and 5,000 controls. The current proposal takes the next logical step by pursuing the most promising findings of our Genome-Wide Association Study (GWAS) to complete the following aims:

Specific Aim #1: Perform deep DNA sequencing of Chr 1q22 among non-Hispanic white and black ICH cases and controls to identify all genomic variation within these regions and test the following:

Hypothesis #1a: Variants strongly associated with ICH risk at 1q22 are either directly causal or in linkage disequilibrium to causal variants that influence ICH risk, and sequencing of these regions will reveal both common and rare variants that exert this causal influence.

Hypothesis #1b: Variants strongly associated with ICH risk at 1q22 will be associated with risk of, or severity of, leukoaraiosis.

Specific Aim #2: Prospectively collect DNA, RNA, and serum on ICH cases and geographic region site-specific controls both at the time of ICH and in the convalescent period. We will perform RNA expression profiling between cases and controls and over time in cases. We will compute expression quantitative trait locus (eQTL) analysis with Single Nucleotide Polymorphisms (SNPs) arising from Aim 1. We will also determine whether alternatively spliced transcripts differ between cases and controls.

Hypothesis #2a: Variation in gene expression or alternatively spliced transcripts affects risk of ICH.

Hypothesis #2b: Variations identified by DNA sequencing will affect gene expression and/or alternatively spliced transcripts that affect risk of ICH.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Resident (6 months or longer) within the recruitment center
* Fulfillment of the criteria for spontaneous ICH
* No evidence of trauma, brain tumor/metastases or infectious processes as a cause of the hemorrhage
* Ability of the patient or legal representative to provide consent for an interview, blood pressure determinations and DNA sampling

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be limited to physician-reviewed cases of people who have had a hemorrhagic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Perform deep DNA sequencing of Chr 1q22 | Ongoing to be completed at the end of June 2021
  Perform deep DNA sequencing of Chr 1q22 among non-Hispanic white and black ICH cases and controls to identify all genomic variation within these regions.

SECONDARY OUTCOMES:
Collect and analyze DNA, RNA, and serum on ICH cases and matched control participants. | Ongoing to be completed at the end of June 2021
  Collect and analyze DNA, RNA, and serum on ICH cases and matched controls both at the time of ICH and in the convalescent period. We will perform RNA expression profiling between cases and controls and over time in cases.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Woo, MD, Principal Investigator — University of Cincinnati
Locations (7):
- United States (7):
  - University of Illinois Chicago, Chicago, Illinois
  - Baptist Health Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woo D, Sauerbeck LR, Kissela BM, Khoury JC, Szaflarski JP, Gebel J, Shukla R, Pancioli AM, Jauch EC, Menon AG, Deka R, Carrozzella JA, Moomaw CJ, Fontaine RN, Broderick JP. Genetic and environmental risk factors for intracerebral hemorrhage: preliminary results of a population-based study. Stroke. 2002 May;33(5):1190-5. doi: 10.1161/01.str.0000014774.88027.22. PMID 11988589
- [Background] Kissela BM, Sauerbeck L, Woo D, Khoury J, Carrozzella J, Pancioli A, Jauch E, Moomaw CJ, Shukla R, Gebel J, Fontaine R, Broderick J. Subarachnoid hemorrhage: a preventable disease with a heritable component. Stroke. 2002 May;33(5):1321-6. doi: 10.1161/01.str.0000014773.57733.3e. PMID 11988610
- [Background] Woo D, Kissela BM, Khoury JC, Sauerbeck LR, Haverbusch MA, Szaflarski JP, Gebel JM, Pancioli AM, Jauch EC, Schneider A, Kleindorfer D, Broderick JP. Hypercholesterolemia, HMG-CoA reductase inhibitors, and risk of intracerebral hemorrhage: a case-control study. Stroke. 2004 Jun;35(6):1360-4. doi: 10.1161/01.STR.0000127786.16612.A4. Epub 2004 Apr 15. PMID 15087556
- [Background] Woo D, Haverbusch M, Sekar P, Kissela B, Khoury J, Schneider A, Kleindorfer D, Szaflarski J, Pancioli A, Jauch E, Moomaw C, Sauerbeck L, Gebel J, Broderick J. Effect of untreated hypertension on hemorrhagic stroke. Stroke. 2004 Jul;35(7):1703-8. doi: 10.1161/01.STR.0000130855.70683.c8. Epub 2004 May 20. PMID 15155969
- [Background] Flaherty ML, Woo D, Haverbusch M, Sekar P, Khoury J, Sauerbeck L, Moomaw CJ, Schneider A, Kissela B, Kleindorfer D, Broderick JP. Racial variations in location and risk of intracerebral hemorrhage. Stroke. 2005 May;36(5):934-7. doi: 10.1161/01.STR.0000160756.72109.95. Epub 2005 Mar 24. PMID 15790947
- [Background] Sauerbeck LR, Khoury JC, Woo D, Kissela BM, Moomaw CJ, Broderick JP. Smoking cessation after stroke: education and its effect on behavior. J Neurosci Nurs. 2005 Dec;37(6):316-9, 325. PMID 16396084
- [Background] Woo D, Kaushal R, Chakraborty R, Woo J, Haverbusch M, Sekar P, Kissela B, Pancioli A, Jauch E, Kleindorfer D, Flaherty M, Schneider A, Khatri P, Sauerbeck L, Khoury J, Deka R, Broderick J. Association of apolipoprotein E4 and haplotypes of the apolipoprotein E gene with lobar intracerebral hemorrhage. Stroke. 2005 Sep;36(9):1874-9. doi: 10.1161/01.STR.0000177891.15082.b9. Epub 2005 Aug 11. PMID 16100021
- [Background] Woo D, Sekar P, Chakraborty R, Haverbusch MA, Flaherty ML, Kissela BM, Kleindorfer D, Schneider A, Khoury J, Sauerbeck LR, Deka R, Broderick JP. Genetic epidemiology of intracerebral hemorrhage. J Stroke Cerebrovasc Dis. 2005 Nov-Dec;14(6):239-43. doi: 10.1016/j.jstrokecerebrovasdis.2005.08.002. PMID 16557295
- [Background] Flaherty ML, Haverbusch M, Kissela B, Kleindorfer D, Schneider A, Sekar P, Moomaw CJ, Sauerbeck L, Broderick JP, Woo D. Perimesencephalic subarachnoid hemorrhage: incidence, risk factors, and outcome. J Stroke Cerebrovasc Dis. 2005 Nov-Dec;14(6):267-71. doi: 10.1016/j.jstrokecerebrovasdis.2005.07.004. PMID 16518463
- [Background] Flaherty ML, Woo D, Haverbusch M, Moomaw CJ, Sekar P, Sauerbeck L, Kissela B, Kleindorfer D, Broderick JP. Potential applicability of recombinant factor VIIa for intracerebral hemorrhage. Stroke. 2005 Dec;36(12):2660-4. doi: 10.1161/01.STR.0000189634.08400.82. Epub 2005 Nov 3. PMID 16269646
- [Background] Woo D, Kaushal R, Kissela B, Sekar P, Wolujewicz M, Pal P, Alwell K, Haverbusch M, Ewing I, Miller R, Kleindorfer D, Flaherty M, Chakraborty R, Deka R, Broderick J. Association of Phosphodiesterase 4D with ischemic stroke: a population-based case-control study. Stroke. 2006 Feb;37(2):371-6. doi: 10.1161/01.STR.0000198843.72824.0a. Epub 2005 Dec 22. PMID 16373644
- [Background] Flaherty ML, Haverbusch M, Sekar P, Kissela B, Kleindorfer D, Moomaw CJ, Sauerbeck L, Schneider A, Broderick JP, Woo D. Long-term mortality after intracerebral hemorrhage. Neurology. 2006 Apr 25;66(8):1182-6. doi: 10.1212/01.wnl.0000208400.08722.7c. PMID 16636234
- [Background] Flaherty ML, Haverbusch M, Sekar P, Kissela BM, Kleindorfer D, Moomaw CJ, Broderick JP, Woo D. Location and outcome of anticoagulant-associated intracerebral hemorrhage. Neurocrit Care. 2006;5(3):197-201. doi: 10.1385/NCC:5:3:197. PMID 17290088
- [Background] Kaushal R, Pal P, Alwell K, Haverbusch M, Flaherty M, Moomaw C, Sekar P, Kissela B, Kleindorfer D, Chakraborty R, Broderick J, Deka R, Woo D. Association of ALOX5AP with ischemic stroke: a population-based case-control study. Hum Genet. 2007 Jun;121(5):601-7. doi: 10.1007/s00439-007-0338-y. Epub 2007 Mar 27. PMID 17387518
- [Background] Eden SV, Morgenstern LB, Sekar P, Moomaw CJ, Haverbusch M, Flaherty ML, Broderick JP, Woo D. The role of race in time to treatment after subarachnoid hemorrhage. Neurosurgery. 2007 May;60(5):837-43; discussion 837-43. doi: 10.1227/01.NEU.0000255451.82483.50. PMID 17460518
- [Background] Kaushal R, Woo D, Pal P, Haverbusch M, Xi H, Moomaw C, Sekar P, Kissela B, Kleindorfer D, Flaherty M, Sauerbeck L, Chakraborty R, Broderick J, Deka R. Subarachnoid hemorrhage: tests of association with apolipoprotein E and elastin genes. BMC Med Genet. 2007 Jul 31;8:49. doi: 10.1186/1471-2350-8-49. PMID 17672902
- [Background] Flaherty ML, Kissela B, Woo D, Kleindorfer D, Alwell K, Sekar P, Moomaw CJ, Haverbusch M, Broderick JP. The increasing incidence of anticoagulant-associated intracerebral hemorrhage. Neurology. 2007 Jan 9;68(2):116-21. doi: 10.1212/01.wnl.0000250340.05202.8b. PMID 17210891
- [Background] Kharofa J, Sekar P, Haverbusch M, Moomaw C, Flaherty M, Kissela B, Broderick J, Woo D. Selective serotonin reuptake inhibitors and risk of hemorrhagic stroke. Stroke. 2007 Nov;38(11):3049-51. doi: 10.1161/STROKEAHA.107.491472. Epub 2007 Sep 27. PMID 17901378